CLINICAL TRIAL: NCT04050007
Title: Effect of a Systematic Preventive Versus Curative Strategy of Fluid Removal on the Weaning of Mechanical Ventilation
Brief Title: Preventive Versus Curative Treatment of Fluid Overload
Acronym: PCT-Fluid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP180559; 2019-A00289-48 (Other: ANSM)
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Preventive initiation of fluid removal
  Interventions: Other: Preventive initiation of fluid removal
- 2 (Other): Curative initiation of fluid removal
  Interventions: Other: Curative initiation of fluid removal

INTERVENTIONS:
Other: Preventive initiation of fluid removal — Preventive initiation of fluid removal will be started right after the randomization with intravenous diuretics according to a predefined algorithm based on the urine output every three hours.
  The weaning process and post extubation preventive strategy will be protocolized based on the last international guidelines
  Arms: 1
Other: Curative initiation of fluid removal — The initiation of fluid removal will be considered by the attending physician only in case of failure to the spontaneous breathing trial with a clinical suspicion of weaning induced pulmonary edema.
  The weaning process and post extubation preventive strategy will be protocolized based on the last international guidelines
  Arms: 2

SUMMARY:
Fluid overload is associated with a poor prognosis in critically ill patients, especially during weaning from mechanical ventilation as it may promote weaning induced pulmonary edema. Previous data suggest that early administration of diuretics ("preventive depletion") could shorten the duration of mechanical ventilation. However, this strategy may expose patients to a risk of metabolic complications. On the other hand, initiating fluid removal only in case of weaning induced pulmonary edema (curative depletion) may reduce the risk of metabolic complications, but prolong the duration of mechanical ventilation. Currently, there is no recommendation for a preventive or curative use of diuretics during weaning. There is therefore an equipoise on the timing of initiation of diuretics during weaning from mechanical ventilation.

DETAILED DESCRIPTION:
Mechanical ventilation is a cornerstone treatment for critically ill patients that is however associated with complications that may alter the prognosis. A major objective is therefore to separate patients from the ventilator as quickly as possible, but without exposing them to the risk of extubation failure. Pulmonary edema is a frequent cause of extubation failure (up to 60% in recent series) and a positive fluid balance has been identified as an important risk factor for extubation failure.

Studies have tested the effect of a conservative strategy regarding the administration of fluids in patients with acute respiratory distress syndrome. This strategy is associated with an improvement in hemodynamic parameters despite an increase in urine output with a negative fluid balance and a significant weight loss as compared to a liberal strategy. The conservative approach also shows a significant improvement in oxygenation with a nonsignificant trend towards a shorter duration of artificial ventilation and ICU stay. During the specific phase of weaning from mechanical ventilation, a randomized trial (BMW trial) demonstrated that a strategy of fluid removal guided by measurement of the plasmatic B-type natriuretic peptide significantly reduced the duration of weaning. Likewise, the interest of obtaining a negative fluid balance through the administration of diuretics in weaning induced pulmonary edema has been established for decades ("curative depletion").

In this context, the hypothesis of the present study is that a preventive and systematic strategy of fluid removal through the use of diuretics initiated just before the weaning phase, as soon as the patients is stabilized would shorten the duration of weaning from mechanical ventilation as compared to a curative strategy of fluid removal, only initiated after a failure of the spontaneous breathing trial associated with weaning induced pulmonary edema.

The design of the study will be a randomized (1:1) controlled trial, open label, with 2 arms, to evaluate the superiority of the preventive strategy.

The weaning process will be protocolized and similar for the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. age>18
2. intubation and mechanical ventilation >= 24 hours
3. cumulative fluid balance judged positive or increase in body weight since admission
4. clinical stability as defined by: 4.1. stable oxygenation (SpO2 ≥ 90 % with FiO2 ≤ 50 % and positive end-expiratory pressure (PEEP) ≤ 8 cm H2O) 4.2. stable hemodynamics (no pressors, no fluid expansion within the last 12 hours) 4.3. stopped or decreased sedation within the last 48 hours and stable neurologic state.

   4.4. temperature >36,0 ◦C and < 39◦C
5. consent signed by the patient or next of kin or emergency procedure

Exclusion Criteria:

1. extracorporal membrane oxygenation
2. pregnancy or breastfeeding
3. allergy to furosemide, sulfamides or spironolactone
4. tracheotomy
5. hydrocephaly
6. acute right ventricle failure
7. cardiac arrest with estimated poor prognosis
8. already enrolled in an interventional study on weaning from mechanical ventilation
9. Guillain Barre, myasthenia crisis
10. planned extubation on the day
11. criteria of clinical stability (as described above) present since more than 24 hours
12. natremia > 150 mEq/L, kaliemia < 3.5 mEq/L, metabolic alkalosis with pH>7.5
13. administration of iodinated contrast within the last 6 hours
14. ongoing or planned use of artificial kidney within the next 48 hours
15. no affiliation to the health insurance system
16. patient under curatorship
17. imprisoned patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Duration of weaning from mechanical ventilation | 28 days
  Time elapsed between the day of randomization and the day of successful extubation (patient alive without reintubation 7 days after extubation)

SECONDARY OUTCOMES:
Percentage of patients with metabolic complications | 28 days
  At least one among hypernatremia (>150 mEq/L), hypokaliemia (<2.5 mEq/L) or kidney injury (KDIGO classification stades 2 et 3)
Percentage of patients with hemodynamic complications | 28 days
  At least one among hypotension with systolic blood pressure <90 mmHg, introduction or increase in vasopressors dose, use of fluid expansion, atrial fibrillation, ventricular fibrillation
Daily and cumulated fluid balance | 28 days
  Difference between fluids intake and output (mL)
Rate of patients who failed the first spontaneous breathing trial | 28 days
  Failure of the first spontaneous breathing trial defined according to international guidelines
Rate of reintubation | 7 days
  Rate of patients who have been reintubated on the basis of predefined criteria (coma, cardiac or respiratory arrest, shock, post extubation acute respiratory distress)
Rate of tracheotomy | 28 days
  Decision of tracheotomy by the attending physician
Percentage of patients with use of unplanned non invasive ventilation (NIV) and high flow nasal cannula (HFNC) oxygen | 7 days
  Decision of use of NIV and HFNC by the attending physician, based on the international guidelines
Ventilator free days | At 14 days and 28 days
  Number of ventilator free days
Total number of days of mechanical ventilation | 28 days
  Number of days from intubation to successful extubation (patient alive without reintubation within 7 days after extubation)
Percentage of patients with ventilator associated pneumonia | 28 days
  as per consensus definition: presence of the 3 criteria:
  * Clinical suspicion (temperature> 38.3 ° C, leukocytosis (> 12000 / mm3) or leukopenia (<4000 / mm3), hypoxemia, auscultatory signs, or septic shock without obvious focus
  * New radiological infiltrate
  * Positive respiratory sampling in culture (quantitative or non-quantitative)
Duration of stay in the ICU | 28 days
  Time elapse from ICU admission to ICU discharge
Duration of stay in the hospital | 28 days
  Time elapse from hospital admission to hospital discharge
Percentage of deaths in the ICU among patients | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- GH Pitié Salpêtrière - Charles Foix, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission Nationale de l'Informatique et des Libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Derived] Dres M, Estellat C, Baudel JL, Beloncle F, Cousty J, Galbois A, Guerin L, Labbe V, Labro G, Lebut J, Mira JP, Prat G, Quenot JP, Dessap A; Reseau Europeen de Recherche en Ventilation Artificielle (REVA) research network. Comparison of a preventive or curative strategy of fluid removal on the weaning of mechanical ventilation: a study protocol for a multicentre randomised open-label parallel-group trial. BMJ Open. 2021 Aug 16;11(8):e048286. doi: 10.1136/bmjopen-2020-048286. PMID 34400454